CLINICAL TRIAL: NCT01263405
Title: Monitoring Chemotherapy Response of Soft Tissue Sarcomas and Osteosarcomas Using Diffuse Optical Spectroscopic Imaging
Status: Completed | Type: Observational
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Bruce Tromberg, PhD., Director, Beckman Laser Institute and Medical Clinic, Professor, Departments of Biomedical Engineering and Surgery, University of California, Irvine
Other Study IDs: 20107852; Department Fund (Other Grant/Funding Number: Department Fund)
Record Dates: First submitted 2010-12-16; First posted 2010-12-20 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Sarcoma
Keywords: Sarcoma
MeSH Terms: conditions — Sarcoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Normal: normal volunteers without sarcoma
- Sarcoma: Sarcoma

SUMMARY:
The purpose of this study is to determine the ability of a specific imaging method, termed Diffuse Optical Spectroscopic Imaging, to provide metabolic and functional information which can be used to predict overall response to preoperative (neoadjuvant) chemotherapy in patients with sarcomas. Sarcoma patients face comparatively poor response rates to chemotherapy and early, non-invasive indications of response could provide physicians with the information necessary to make evidence-based changes in treatment strategies. Patients who do not demonstrate early signs of response would be spared the unnecessary side-effects of an ineffective chemotherapy regimen, and could either be switched to a different regimen or undergo surgery

DETAILED DESCRIPTION:
In this study we plan to measure bone and soft tissue sarcoma patients using Diffuse Optical Spectroscopic Imaging to determine if analogous markers of response exist for these patients. The first aim of this study is to measure normal volunteers using Diffuse Optical Spectroscopic Imaging in the anatomic regions where sarcomas typically occur such as the extremities. This will provide normal optical properties with which to compare sarcoma measurements. The second aim of this study is to determine the feasibility of measuring sarcoma patients with Diffuse Optical Spectroscopic Imaging. Since the optical properties of sarcoma tissue will likely be different from breast tumor tissue, we will measure a small cohort of patients at baseline (before treatment) to determine typical optical properties and make any necessary instrument adjustments. The third aim of the study will involve measuring sarcoma patients using Diffuse Optical Spectroscopic Imaging at multiple timepoints during their treatment including at baseline, during their first week of neoadjuvant chemotherapy, at the midpoint of therapy, and before surgical resection. Additionally, some patients may be measured during their chemotherapy infusions as this timepoint has shown promising preliminary data in breast cancer patients. Diffuse Optical Spectroscopic Imaging measurements will be analyzed and compared to overall chemotherapy response determined by pathology. Additionally, DOSI measurements will be compared to clinical MRI (or FDG PET/CT) measurements performed at baseline and at posttreatment prior to surgery according to RECIST/PERCIST criteria. Tumor volume reduction (or tumor metabolic change) during chemotherapy will be compared to Diffuse Optical Spectroscopic Imaging measurements. Finally, as a fourth study aim, biopsy specimens from patients will be analyzed by immunohistochemistry for metabolic, proliferative, and necrotic markers. These markers will be correlated with optical markers to help further understand the how DOSI can inform physicians about the tumor biology of sarcomas.

ELIGIBILITY:
Inclusion Criteria:

* Any subjects with no current or previous history of sarcoma are eligible to be a normal volunteer
* Any subject with a sarcoma neoplasm is eligible to be measured for aim 2 of the study
* Only patients undergoing neoadjuvant chemotherapy for sarcoma are eligible for Aim 3 of the study

Exclusion Criteria:

* Age less that 18 year old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic and community sample
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2010-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Monitoring Chemotherapy Response of Soft Tissue Sarcomas and Osteosarcomas | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Tromberg, PhD, Principal Investigator — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute, Irvine, California, United States